CLINICAL TRIAL: NCT01525654
Title: Rheumatoid Arthritis Patient-to-Patient Connection Program
Brief Title: Patient Rheumatoid Arthritis Social Support Study
Acronym: PARASS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ran out of funding
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Nancy Shadick, Associate Professor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2006P000795
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; peer support; self-efficacy; medication adherence
MeSH Terms: conditions — Arthritis, Rheumatoid; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partners (Active Comparator): Patients who are matched with support partners and have a billing diagnosis of RA (714.0) or seronegative inflammatory arthritis who are enrolled in the Brigham and Women's Rheumatoid Arthritis Sequential Study (BRASS) or the Patient-Centered Outcomes Initiative (PACO)
  Interventions: Behavioral: Peer Support Program
- Controls (No Intervention): Controls will be BRASS patients who continue to receive regular care without being matched with a peer support partner.

INTERVENTIONS:
Behavioral: Peer Support Program — Partners, are interested in having a support person to talk with while others. Coaches initiate contact, usually via phone but can use email or face to face, with their Partner. During this initial contact, partners determine how often to speak up to a total of 6 months. Peer Support discussions focus on sharing information, education, support related to living with RA.
  Arms: Partners

SUMMARY:
The goal of PARASS is to develop a network of increased social support for Rheumatoid Arthritis (RA) patients that will improve patient outcomes and further promote understanding of RA among physicians and patients in the clinic community. This will be accomplished with the development and implementation of Buddy pairing and one -on- one informational support to be called Patient-to-Patient Connection.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic disabling disease that affects nearly 1% of the U. S. population [1]. The illness causes destruction of joint cartilage and erosion of adjacent bone, leading to joint replacement as well as extra-articular disease including cardiopulmonary manifestations, vasculitis, gastrointestinal and infectious complications [2]. Many patients with RA over time suffer progressive disability [3, 4], pain [5], work loss [3, 6], substantial health care costs [7], and premature mortality [8]. The current treatment of RA results in only modest improvements in functional status and many patients progress to chronic disability. Treatment is focused on ameliorating symptoms and halting disease progression as early as possible to prevent joint damage and functional decline.

Research has shown that while patient response to different medications may vary, those with chronic illness universally require social support and human empathy to achieve the best physical and emotional outcomes. From the 2006 PACO focus groups, we learned that RA patients' greatest concern was social isolation, that almost all had never talked with another person with RA, and that they feel alone dealing with the challenges of the disease. Psychosocial support is a seminal aspect of disease management since interpersonal relationships are often affected by the fatigue and physical disability of the disease and self-efficacy by the resulting loss of independence. The purpose of this study is to further patient care by providing social support services to better arthritis outcomes and patient satisfaction. In this pilot initiative called PARASS Patient-to-Patient Connection, patients will be able to connect with fellow patients who have similar concerns and fears and can find empathy and understanding based on personal experience. Buddy systems matching patients with similar needs or interests have been successful in addiction rehabilitation and oncology treatment, and group sessions have long been used as teaching and support tools in diabetes management. Rheumatology, however, has to date focused largely on providing patients with tools to improve the more physical manifestations of pain, swelling and fatigue. Furthermore, efforts to enhance self efficacy through leader initiated self help courses have not produced expected improvements in clinical outcomes. The purpose of this initiative is to develop a novel method of patient empowerment using peer support in order to better arthritis outcomes and patient satisfaction. To our knowledge, no rheumatology clinics in the United States have developed or instituted organized programs for peer social support or group informational discussion.

The goal of PARASS is to develop a network of increased social support for Rheumatoid Arthritis (RA) patients that will improve patient outcomes and further promote understanding of RA among physicians and patients in the clinic community. This will be accomplished with the development and implementation of a "buddy pairing" program called Patient-to-Patient Connection.

ELIGIBILITY:
Inclusion Criteria:

* billing diagnosis of rheumatoid arthritis (714.0) or seronegative inflammatory arthritis or a member of the BRASS and PACO studies at Brigham and Women's Hospital

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
change in functional status | baseline and 6 months
  functional status is measured by the Multi Dimensional Health Assessment Questionnaire doing scale and flare activity
change in medication adherence | baseline and 6 months
  assessed with the Adherence Barrier Survey-20 medication adherence questionnaire

SECONDARY OUTCOMES:
change in self-efficacy | baseline and 6 months
  assessed using the Arthritis Self-Efficacy Scale
change in fatigue | baseline and 6 months
  assessed by the Multi Dimensional Health Assessment Questionnaire Visual Analog Scale fatigue question
change in pain | baseline and 6 months
  assessed by the Multi Dimensional Health Assessment Questionnaire Visual Analog Scale pain question

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Linos A, Worthington JW, O'Fallon WM, Kurland LT. The epidemiology of rheumatoid arthritis in Rochester, Minnesota: a study of incidence, prevalence, and mortality. Am J Epidemiol. 1980 Jan;111(1):87-98. doi: 10.1093/oxfordjournals.aje.a112878. PMID 7352462
- [Background] Pincus T, Callahan LF, Sale WG, Brooks AL, Payne LE, Vaughn WK. Severe functional declines, work disability, and increased mortality in seventy-five rheumatoid arthritis patients studied over nine years. Arthritis Rheum. 1984 Aug;27(8):864-72. doi: 10.1002/art.1780270805. PMID 6431998
- [Background] Sherrer YS, Bloch DA, Mitchell DM, Young DY, Fries JF. The development of disability in rheumatoid arthritis. Arthritis Rheum. 1986 Apr;29(4):494-500. doi: 10.1002/art.1780290406. PMID 3707627
- [Background] Callahan LF, Brooks RH, Summey JA, Pincus T. Quantitative pain assessment for routine care of rheumatoid arthritis patients, using a pain scale based on activities of daily living and a visual analog pain scale. Arthritis Rheum. 1987 Jun;30(6):630-6. doi: 10.1002/art.1780300605. PMID 3606681
- [Background] Yelin E, Meenan R, Nevitt M, Epstein W. Work disability in rheumatoid arthritis: effects of disease, social, and work factors. Ann Intern Med. 1980 Oct;93(4):551-6. doi: 10.7326/0003-4819-93-4-551. PMID 7436187
- [Background] Meenan RF, Yelin EH, Henke CJ, Curtis DL, Epstein WV. The costs of rheumatoid arthritis. A patient-oriented study of chronic disease costs. Arthritis Rheum. 1978 Sep-Oct;21(7):827-33. doi: 10.1002/art.1780210714. PMID 100122
- [Background] Pincus T, Brooks RH, Callahan LF. Prediction of long-term mortality in patients with rheumatoid arthritis according to simple questionnaire and joint count measures. Ann Intern Med. 1994 Jan 1;120(1):26-34. doi: 10.7326/0003-4819-120-1-199401010-00005. PMID 8250453
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Hahn SR, Park J, Skinner EP, Yu-Isenberg KS, Weaver MB, Crawford B, Flowers PW. Development of the ASK-20 adherence barrier survey. Curr Med Res Opin. 2008 Jul;24(7):2127-38. doi: 10.1185/03007990802174769. Epub 2008 Jun 12. PMID 18554431
- [Background] Harris, E.D., Rheumatoid arthritis. 1997, Philadelphia: Saunders. xxiii, 433.
- See also: Related Info — http://parassstudy.org